CLINICAL TRIAL: NCT06074042
Title: The Clinical Characteristics, Treatment and Prognosis of Tuberculosis-associated Chronic Obstructive Pulmonary Disease in China: A Multicenter Prospective Cohort Study
Brief Title: The Clinical Characteristics, Treatment and Prognosis of Tuberculosis-associated COPD
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); First Hospital of China Medical University (Other); West China Hospital (Other); Shanxi Bethune Hospital (Other); Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Principal Investigator, Liang Ying, Peking University Third Hospital, Peking University Third Hospital
Other Study IDs: M2023573
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease (COPD); acute exacerbation of COPD; pulmonary tuberculosis; phenotype
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tuberculosis-associated COPD: COPD patient who meets any of the following criteria is diagnosed as tuberculosis-associated COPD:
  1. previously definite pulmonary tuberculosis and ever receiving standard antituberculosis therapy;
  2. previously suspected pulmonary tuberculosis and having typical radiological findings consistent with tuberculosis sequelae;
  3. no definite history of pulmonary tuberculosis but having positive T-SPOT.TB test accompanied with typical radiological findings consistent with tuberculosis sequelae.
  Interventions: Other: previous pulmonary tuberculosis
- non-tuberculosis associated COPD: COPD patient in whom neither medical history nor chest CT indicates evidence of pulmonary tuberculosis is diagnosed as non-tuberculosis associated COPD.

INTERVENTIONS:
Other: previous pulmonary tuberculosis — Previous pulmonary tuberculosis is comprehensively evaluated by the self-reported medical history, T-SPOT.TB test and radiological findings.
  Groups: tuberculosis-associated COPD

SUMMARY:
Chronic obstructive pulmonary disease (COPD) still imposes a substantial health and economic burden worldwide. Pulmonary tuberculosis has been confirmed as an important risk factor for COPD and this specific phenotype is thereby named as "tuberculosis-associated COPD". Although it is a generally accepted concept, several relevant problems need to be addressed, including how to define this phenotype more precisely, what the clinical characteristics and prognosis are as well as which kind of pharmacologic intervention is optimal.

In this study, tuberculosis-associated COPD patients (study group) and non-tuberculosis associated COPD patients (control group) are recruited. After collecting baseline information of participants, the investigators arrange for participants to follow up in the outpatient for reassessment with a scheduled interval of 6 months, which lasts for 1 year. Primary outcome of this study is the frequency of moderate/severe acute exacerbation of COPD during the follow-up of 12 months. By conducting a multicenter prospective cohort study in China, the researchers intend to investigate the clinical characteristics and prognostic predictors, explore plausible therapeutic regimens and promote precise diagnosis and treatment for tuberculosis-associated COPD.

DETAILED DESCRIPTION:
A nationwide, multicenter, prospective, observational cohort study enrolling consecutive tuberculosis-associated COPD patients (study group) and non-tuberculosis associated COPD patients (control group) is designed to conduct across mainland China, in which a total of 7 tertiary hospitals will participate. Stable COPD patients meeting the criteria will be allocated into "tuberculosis-associated COPD group" or "non-tuberculosis associated COPD group" according to the medical history, T cell spot test for tuberculosis infection (T-SPOT.TB) and chest computed tomography (CT) sign. Baseline information of the participants will be collected, including the following items:

* Demographic data. Age, sex, ethnicity, height, weight, residential address, education level and annual household income will be collected;
* Smoking history and medical history associated with pulmonary tuberculosis and COPD;
* Therapeutic regimens for COPD;
* Respiratory symptoms evaluated by the COPD Assessment Test (CAT) score, the modified Medical Research Council (mMRC) dyspnea scale and St George's Respiratory Questionnaire for COPD patients (SGRQ-C);
* Blood routine examination and T-SPOT.TB;
* Lung function. Pre-bronchodilator and post-bronchodilator spirometry function and diffusing capacity are assessed;
* Chest CT. Radiological findings about tuberculosis sequelae include calcification, fibrotic lesions, dense nodules, cavitation or pleural scarring. Severity of emphysema is evaluated by using Goddard score. Severity and extent of bronchiectasis are evaluated by using Smith score and Bhalla score, respectively.

All participants will be prospectively followed up for at least one year in the outpatient of each affiliated hospitals with an interval of 6 months. Alteration of respiratory symptom, lung function and blood routine examination, therapeutic regimen, chest CT, frequency of exacerbation and hospitalization as well as total expenditure associated with COPD will be reevaluated and recorded. The frequency of moderate/severe acute exacerbation of COPD during the follow-up of 12 months is the primary outcome.

Main objectives of this study are about the following aspects:

1. Elucidate the clinical characteristics, progression and prognosis of tuberculosis-associated COPD.
2. Evaluate the relationship between different drug regimens and the prognosis of tuberculosis-associated COPD, as well as recurrence or deterioration of pulmonary tuberculosis, serving to the personalized medical management.
3. Optimize the definition of tuberculosis-associated COPD.

ELIGIBILITY:
Inclusion Criteria:

* patients who have dyspnea, chronic cough or sputum production and have definite airflow limitation with a post-bronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) <0.7;
* in stable condition;
* aged 35 years or older

Exclusion Criteria:

* bronchiectasis, asthma or any other obstructive pulmonary diseases;
* pneumonia or active tuberculosis;
* severe hepatic or renal insufficiency;
* lung cancer or other advanced malignancies;
* acquired immune deficiency due to HIV or chemotherapy;
* severe trauma, operation or stress status in the past one month;
* severe cognitive dysfunction;
* unwilling to provide informed consent

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from seven hospitals distributed in 6 different provinces of China.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the frequency of moderate/severe acute exacerbation of COPD during the follow-up of 12 months | Through study completion, an average of 1 year
  Exacerbations of COPD are defined as sustained increase of respiratory symptoms characterized by dyspnea and/or cough and sputum. Classification of severity of COPD exacerbations is as followed:
  * Mild. Only monotherapy of short-acting bronchodilator is prescribed for treatment;
  * Moderate. Short-acting bronchodilator and antibacterial agents are prescribed combined with oral glucocorticoids or not;
  * Severe. Hospitalization or admission to intend care unit (ICU) is required.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liang, M.D., Principal Investigator — Peking University Third Hhospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No